CLINICAL TRIAL: NCT02824887
Title: A Prospective Cohort Study of Electroacupuncture Deep Needling Protrusion of Lumbar Intervertebral Disc the Five Acupoints in the Treatment of Lumbar Disc Herniation
Brief Title: Deep Needling Protrusion of Lumbar Intervertebral Disc the Five Acupoints
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated Hospital of Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhao Jian Xin, Chief physician, The Third Affiliated Hospital of Beijing University of Chinese Medicine
Other Study IDs: 40083459-X
Record Dates: First submitted 2016-06-05; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Protrusion of Lumbar Intervertebral Disc
Keywords: Electroacupuncture; Deep needling; Lumbar disc herniation five points; Long term effect; Prospective cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed group: Long term curative effect of electroacupuncture treatment of lumbar intervertebral disc herniation in exposure group
  Interventions: Other: Electro-acupuncture
- control group: Long term efficacy of conventional treatment of lumbar disc herniation in the control group
  Interventions: Other: Conventional treatment of Western Medicine

INTERVENTIONS:
Other: Electro-acupuncture — Electro acupuncture deep needling protrusion of lumbar intervertebral disc the five acupoints
  Groups: Exposed group
Other: Conventional treatment of Western Medicine — Routine non operative treatment of Western Medicine
  Groups: control group

SUMMARY:
Compare the curative effects of electroacupuncture deep needling difference in efficacy of the conservative treatment for lumbar five point therapy and routine western medicine, to explore the efficacy and superiority, open a new way for the treatment of lumbar disc herniation.Through a comparative analysis of the data on the efficacy of different TCM Syndrome Types in the subgroup of patients with, to explore the effect of Electroacupuncture of deep needling and five lumbar acupoint therapy is most suitable for the TCM syndrome type.Through follow-up, patients in the two groups moment condition and the survival of the state was evaluated, explore the effect of electroacupuncture deep needling the long-term effects of five lumbar acupoint therapy for treatment of lumbar disc herniation and factors that may influence the recurrence of symptoms.

DETAILED DESCRIPTION:
Beijing and North China area is lumbar protrusion of the intervertebral disc is the most prevalent area, much due to white-collar workers movement amount is small, the long-term bad posture, or do not move for a long time does not accept the ultraviolet radiation due to osteoporosis. The lumbar disc herniation in young people in a year of rapid growth trend, serious illness and severe low back pain even cannot move and accompanied by paralysis of the legs, hair is cool, weakness, intermittent claudication even muscle atrophy and neurological dysfunction, and so on. Some of them have already caused the degeneration of intervertebral disc or the phenomenon of aging. Recent studies show that only 10% - 20% of the lumbar disc herniation patients need surgical treatment, for does not have the surgery patients with, choice of a curative effect, quick effect and side effects of small, simple conservative treatment methods become many lumbar intervertebral disc herniation were urgent needs.Electroacupuncture and deeply needling five lumbar acupoint therapy is the person in charge of the project after more than 20 years of clinical experience put forward the innovation specific therapy is a novel method for the treatment and prognosis of lumbar protrusion of the intervertebral disc to carry out the innovative clinical research applications, both at home and abroad there is no precedent. The project team through a small range of clinical research and literature research have confirmed the efficacy of electro acupuncture treatment of lumbar disc herniation is reliable, but the long-term efficacy of acupuncture therapy has not been carried out. Therefore, combined with the cohort study of conventional medical practice without human intervention, the results of the study more in line with the actual advantages of the design prospective cohort study. Through long-term follow-up, with a large number of clinical evidence of electroacupuncture deep needling five lumbar acupoint therapy for treatment of lumbar disc herniation with conventional western medicine conservative treatment when compared to the differences in efficacy, treatment, recurrence rate, and to explore the long-term effect of lumbar disc herniation recurrence factors and this kind of therapy in the treatment of lumbar disc herniation.This project involved deep needling lumbar five points and long-term follow-up of the key contents and fit the lumbar disc herniation rate high, and recurrent episodes of the characteristics of the course of lingering, represents a concern in modern medical disease curative effect at the same time pay more attention to the development direction of the prognosis of the disease, with good prospects for clinical application. After 1 year, 175 patients visit and follow up the formation of the research results, will be able to EA deep needling lumbar five point therapy to provide high quality clinical evidence, and gradually formed this kind of special treatment as the core characteristics of traditional Chinese medicine treatment pattern, promote the hospital in clinical characteristics and advantages of the party to the development. And in order to attract patients with indications, the amplification of the unit's outpatient volume, to achieve indirect economic benefits. From the social point of view, this study explore drawn about the clinical results and the research process of the patients for rehabilitation guidance, will be of direct benefit to the patient's path choice, for long-term efficacy and prognosis of diseases and lay a good foundation, reduce disease recurrence to help patients to relieve pain, shorten the course of disease, saving the cost of medical treatment. At the same time, a large number of clinical cases of the subject group will be used to establish a database of patients with lumbar disc herniation, which is convenient for the retrospective study in the future. This study through the practice of training training a group with high data acquisition and doctor-patient communication skills and master the characteristics and effective treatment method for the researchers, will also become the support project subject to bear the backbone of the sustainable development.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the criteria for the diagnosis
2. The people whose age are between 18 to 75 years old.
3. Course of no more than 20 years.
4. TCM syndrome type belong to blood stasis, cold dampness syndrome, hot and humid, liver and kidney deficiency license.
5. Pathological classification belongs to unilateral disc herniation or bilateral slipped disc.
6. Signed informed consent will be.

Exclusion Criteria:

1. Patients with severe lumbar disc herniation with surgical indications.
2. Complicated by severe developmental spinal stenosis or other severe malformations.
3. Weak constitution, or pregnant women, etc.
4. Suffers from severe heart disease, high blood pressure, liver and kidney disease patients.
5. Skin damage, ulceration or skin disease.
6. Has a bleeding tendency in patients with hematologic diseases.
7. Psychiatric patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar disc herniation from department of acupuncture and moxibustion in Third affiliated hospital of Beijing university of Chinese medicine
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
JOA | through study completion, an average of 13 months；before treatment，after the sixth treatment，after 3 months of treatment ，after 6 months of treatment ，after 1 year of treatment
VAS | through study completion, an average of 13 months；before treatment，after the sixth treatment，after 3 months of treatment ，after 6 months of treatment ，after 1 year of treatment
SF-36 quality of life questionnaire | Follow-up after treatment，period of about a year
Oswestry functional disorder questionnaire | Follow-up after treatment，period of about a year

SECONDARY OUTCOMES:
Patient satisfaction rating scale | Follow-up after treatment，period of about a year
Influencing factors questionnaire | Follow-up after treatment，period of about a year

CONTACTS AND LOCATIONS:
Overall Officials: Guo Sheng Jun, undergraduate, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Wang Yi Li, undergraduate, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Li Dan, doctor, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Zhou Pei Juan, master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Song Jia Shan, doctor, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Liu Ya Ru, master, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Song Yu Hui, undergraduate, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Li Zhao Qiang, undergraduate, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine; Zhang Hai Xia, undergraduate, Principal Investigator — The Third Affiliated Hospital of Beijing University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided